CLINICAL TRIAL: NCT05038072
Title: Suprachoroidal Triamcinolone Acetonide for the Treatment of Macular Edema Associated With Retinal Vein Occlusion: A Pilot Study
Brief Title: The Use of Suprachoroidal Triamcinolone Acetonide to Treat Macular Edema in Retinal Vein Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UDMS-Opthal-01-2021
Record Dates: First submitted 2021-08-24; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Macular Edema; Retinal Vein Occlusion
Keywords: Macular Edema; Retinal Vein Occlusion; Suprachoroidal Space; Triamcinolone Acetonide; RVO; ME
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion; Choroidal Effusions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4 mg Triamcinolone Acetonide (TA)/ Suprachoriodal Injection (Experimental): Suprachoroidal injection of 4 mg in 100 μL of TA was administered as a single injection.
  Interventions: Drug: suprachoroidal injection of Triamcinolone Acetonide.

INTERVENTIONS:
Drug: suprachoroidal injection of Triamcinolone Acetonide. — 4 mg /0.1 ml TA was injected in the SCS using an individualized microinjector according to scleral thickness measured by anterior segment OCT (AS-OCT) at the injection point (4 mm from the limbus in the inferotemporal quadrant).
  Other Names: SCTA

SUMMARY:
This prospective non-randomized open-label interventional study aimed to evaluate feasibility in regard to potential efficacy and safety of triamcinolone acetonide (TA) injected in the suprachoroidal space (SCS) as a promising therapeutic route that provides a better bioavailability, longer sustained duration of action, and thus improved patients' compliance for the treatment of macular edema due to retinal vein occlusion (RVO).

DETAILED DESCRIPTION:
Management of Macular Edema (ME) associated with Retinal Vein Occlusion (RVO) still poses a therapeutic challenge taking into account its complicated etiopathogenesis. Despite improved visual and anatomical outcomes achieved by intravitreal injections of antiangiogenics and steroids, these treatments are still associated with non-responders, tachyphylaxis, rebound phenomenon, high re-injection, and adverse events rates, which underscore the importance of addressing new approaches to formulate treatment strategies.

Delivery of therapeutic agents into the suprachoroidal space (SCS) provides a novel alternative approach that has theoretical appeal, as it dominantly targets chorioretinal tissues with the posterior and circumferential spread of the drug administered while relatively sparing the unaffected anterior segment of the eye and the vitreous chamber, thus minimizing risks associated with off-target effects, which potentiates safety. This was well translated in preclinical and clinical studies through microinjector, which has been shown to provide a safe, minimally invasive, and reliable method of targeting SCS. In addition, sustained duration and favorable pharmacokinetics have been observed for small molecule suspensions including Triamcinolone Acetonide (TA), with the potential to reduce treatment burden.

ELIGIBILITY:
Inclusion Criteria:

1. Male or nonpregnant female patients >18 years of age.
2. Has a clinical diagnosis of Retinal Vein Occlusion (RVO) in the study eye.
3. Best-Corrected Visual Acuity (BCVA) in Early Treatment Diabetic Retinopathy Study (ETDRS) letter score ≥ 20 (20/400 Snellen equivalent), and ≤75 in the study eye (20/32 Snellen equivalent).
4. Central Subfield Thickness (CST) ≥310 microns measured by Spectral Domain Optical Coherence Tomography (SD-OCT) in the study eye.

Exclusion Criteria:

1. Intravitreal (IVT) injection of anti-VEGF: Bevacizumab (Avastin; Genentech, South San Francisco, CA, USA/Roche, Basel, Switzerland) or ranibizumab (Lucentis; Genentech Inc., South San Francisco, CA, USA) within 1 month and aflibercept (Eylea®; Regeneron Pharmaceuticals Inc., Tarrytown, NY, USA, and Bayer HealthCare Pharmaceuticals, Berlin, Germany) within 2 months in the study eye.
2. Intraocular or periocular corticosteroid injection within 3 months, dexamethasone implant (Ozurdex, Allergan, Dublin, Ireland) within 6 months, Retisert (Bausch and Lomb, Bridge water, NJ) within 1 year, or fluocinolone acetonide implant (Iluvien, Alimera Sciences, Alpharetta, GA) within 3 years in the study eye.
3. Macular laser photocoagulation treatment in the study eye.
4. Topical ophthalmic nonsteroidal anti-inflammatory drugs in the study eye within a month.
5. Any significant media opacity that could hinder the evaluation of the retina or ocular condition causing decreased vision other than RVO.
6. IOP >22 mm Hg, or history of steroid-induced ocular hypertension; uncontrolled glaucoma.
7. Past vitreoretinal or glaucoma surgery in the study eye.
8. Uncontrolled systemic disease that could hinder follow-up, immunodeficiency, or any other systemic contraindication for steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2020-11-22 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with BCVA gain≥ 15 Letters at 3 months | 3 months after injection
  Percentage of participants with ≥ 15 letter Improvement from Baseline Best corrected visual acuity (BCVA) using Early Treatment of Diabetic Retinopathy Study (ETDRS) visual acuity score: BCVA refers to the measurement of the best possible vision that can be achieved following refraction. BCVA was assessed using a Snellen chart. The resultant measures were converted to Early Treatment of Diabetic Retinopathy Study ETDRS letter score. An increase from the pre-treatment state in BCVA of 15 letters or more represents a clinically meaningful improvement.
Percentage of participants with IOP ≥20 mm Hg at 3 months | 3 months after injection
  Intraocular pressure (IOP) is the fluid pressure inside the eye. Tonometry is the method that eye care professionals use to determine this. Tonometers in this study were calibrated to measure pressure in millimeters of mercury.

SECONDARY OUTCOMES:
Change in the BCVA | 1 week, 1 month, 2 months and 3 months after injection.
  Best corrected visual acuity (BCVA) refers to the measurement of the best possible vision that can be achieved following refraction. BCVA was assessed using a Snellen chart. The resultant measures were converted to ETDRS letter score. A positive change from baseline value represents an improvement in vision.
Change in the CST | 1 week, 1 month, 2 months and 3 months after injection.
  Central subfield thickness (CST) is a diagnostic measurement used in identifying the presence of edema in the circular area 1 mm in diameter centered around the fovea. CST was measured using spectral domain optical coherence tomography (SD-OCT) (Heidelberg Spectralis; Heidelberg Engineering, Germany). A negative change from baseline value represents a reduction in macular edema.
Change in the Proportion of Participants with CST ≤ 320 μ | 1 week, 1 month, 2 months and 3 months after injection.
  Central subfield thickness (CST) is the average macular thickness in the central circular area 1 mm in diameter centered around the fovea and is a diagnostic measurement applied to diagnose macular edema. CST was measured using spectral domain optical coherence tomography (SD-OCT) (Heidelberg Spectralis; Heidelberg Engineering, Germany).
Change in the Percentage of Reduction in Excess Foveal Thickness (EFT) | 1 week, 1 month, 2 months and 3 months after injection.
  Excess Foveal Thickness (EFT) was estimated by subtracting 310 µ from the central subfield thickness (CST). CST was measured using spectral domain optical coherence tomography (SD-OCT) (Heidelberg Spectralis; Heidelberg Engineering, Germany).
Change in the Serious Treatment-Emergent Adverse Events (S-TEAEs) | 1 week, 1 month, 2 months and 3 months after injection.
  Number of patients with Serious Treatment-Emergent Adverse Events (S-TEAEs): A treatment-emergent adverse event (TEAE) is the development of an undesirable medical condition or the worsening of a preexisting medical condition either in intensity or frequency after exposure to a pharmaceutical product. Ophthalmic Serious TEAEs include Endophthalmitis, intraocular inflammation, vitreal hemorrhage, retinal tear and Rhegmatogenous retinal detachment.
  These Adverse Events were evaluated through anterior and posterior segments examination using slit lamp biomicroscopy and indirect ophthalmoscopy.
Change in the IOP | 1 week, 1 month, 2 months and 3 months after injection.
  Intraocular pressure (IOP) is the fluid pressure inside the eye. Tonometry is the method that eye care professionals use to determine this. Tonometers in this study were calibrated to measure pressure in millimeters of mercury.

CONTACTS AND LOCATIONS:
Overall Officials: Boushra M Ali, M.D., MRCSEd, Principal Investigator — Resident , Department of Ophthalmology, Faculty of Medicine, Damascus University; Arwa M Azmeh, Ph.D., Study Chair — Professor of Ophthalmology, Department of Ophthalmology, Faculty of Medicine, Damascus University
Locations (1):
- Al Mouwasat University Hospital, Department of Ophthalmology, Damascus, Syria

REFERENCES:
- [Background] Campochiaro PA, Sophie R, Pearlman J, Brown DM, Boyer DS, Heier JS, Marcus DM, Feiner L, Patel A; RETAIN Study Group. Long-term outcomes in patients with retinal vein occlusion treated with ranibizumab: the RETAIN study. Ophthalmology. 2014 Jan;121(1):209-219. doi: 10.1016/j.ophtha.2013.08.038. Epub 2013 Oct 7. PMID 24112944
- [Background] Spooner K, Fraser-Bell S, Hong T, Chang AA. Five-year outcomes of retinal vein occlusion treated with vascular endothelial growth factor inhibitors. BMJ Open Ophthalmol. 2019 Mar 29;4(1):e000249. doi: 10.1136/bmjophth-2018-000249. eCollection 2019. PMID 30997407
- [Background] Ciulla T, Pollack JS, Williams DF. Visual acuity outcomes and anti-VEGF therapy intensity in macular oedema due to retinal vein occlusion: a real-world analysis of 15 613 patient eyes. Br J Ophthalmol. 2021 Dec;105(12):1696-1704. doi: 10.1136/bjophthalmol-2020-317337. Epub 2020 Oct 14. PMID 33055088
- [Background] Moisseiev E, Loewenstein A, Yiu G. The suprachoroidal space: from potential space to a space with potential. Clin Ophthalmol. 2016 Jan 25;10:173-8. doi: 10.2147/OPTH.S89784. eCollection 2016. PMID 26869750
- [Background] Hancock SE, Wan CR, Fisher NE, Andino RV, Ciulla TA. Biomechanics of suprachoroidal drug delivery: From benchtop to clinical investigation in ocular therapies. Expert Opin Drug Deliv. 2021 Jun;18(6):777-788. doi: 10.1080/17425247.2021.1867532. Epub 2021 Jan 3. PMID 33393391
- [Background] Wan CR, Muya L, Kansara V, Ciulla TA. Suprachoroidal Delivery of Small Molecules, Nanoparticles, Gene and Cell Therapies for Ocular Diseases. Pharmaceutics. 2021 Feb 22;13(2):288. doi: 10.3390/pharmaceutics13020288. PMID 33671815
- [Background] Habot-Wilner Z, Noronha G, Wykoff CC. Suprachoroidally injected pharmacological agents for the treatment of chorio-retinal diseases: a targeted approach. Acta Ophthalmol. 2019 Aug;97(5):460-472. doi: 10.1111/aos.14042. Epub 2019 Jan 31. PMID 30702218
- [Background] Chiang B, Jung JH, Prausnitz MR. The suprachoroidal space as a route of administration to the posterior segment of the eye. Adv Drug Deliv Rev. 2018 Feb 15;126:58-66. doi: 10.1016/j.addr.2018.03.001. Epub 2018 Mar 12. PMID 29545195
- [Background] Campochiaro PA, Wykoff CC, Brown DM, Boyer DS, Barakat M, Taraborelli D, Noronha G; Tanzanite Study Group. Suprachoroidal Triamcinolone Acetonide for Retinal Vein Occlusion: Results of the Tanzanite Study. Ophthalmol Retina. 2018 Apr;2(4):320-328. doi: 10.1016/j.oret.2017.07.013. Epub 2017 Sep 29. PMID 31047241
- [Background] Wan CR, Kapik B, Wykoff CC, Henry CR, Barakat MR, Shah M, Andino RV, Ciulla TA. Clinical Characterization of Suprachoroidal Injection Procedure Utilizing a Microinjector across Three Retinal Disorders. Transl Vis Sci Technol. 2020 Oct 22;9(11):27. doi: 10.1167/tvst.9.11.27. eCollection 2020 Oct. PMID 33150052
- [Derived] Ali BM, Azmeh AM, Alhalabi NM. Suprachoroidal triamcinolone acetonide for the treatment of macular edema associated with retinal vein occlusion: a pilot study. BMC Ophthalmol. 2023 Feb 10;23(1):60. doi: 10.1186/s12886-023-02808-5. PMID 36765332